CLINICAL TRIAL: NCT06997744
Title: Comparative Effects of 2Hz Versus 100Hz Transcutaneous Electrical Nerve Stimulation on Upper Limb Motor Function Post-Stroke: Design and Rationale for a Randomized Trial
Brief Title: TENS for Limb Function in Stroke: Design and Rationale for a Randomized Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHENGNING Song (Other)
Responsible Party: Sponsor-Investigator, CHENGNING Song, Doctor, Shenzhen Baoan District Fuyong People's Hospital
Organization: Shenzhen Baoan District Fuyong People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY-2025-111
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 2Hz TENS Group (Experimental)
  Interventions: Device: Low-frequency(2HZ) TENS
- 100Hz TENS Group (Experimental)
  Interventions: Device: High-frequency(100HZ) TENS
- Placebo TENS Group (Placebo Comparator)
  Interventions: Device: Placebo TENS
- No-treatment Control Group (No Intervention)

INTERVENTIONS:
Device: Low-frequency(2HZ) TENS — Participants receive transcutaneous electrical nerve stimulation (TENS) at a frequency of 2Hz. The stimulation is delivered using surface electrodes placed on the affected upper limb. Each session lasts 30 minutes and is conducted three times per week for a total of 8 weeks. Intensity is gradually increased from 1 mA to 3 mA during each session.
  Arms: 2Hz TENS Group
Device: High-frequency(100HZ) TENS — Participants receive TENS at a frequency of 100Hz using the same electrode placement and schedule as the 2Hz group. Sessions last 30 minutes, three times weekly for 8 weeks, with intensity increasing from 1 mA to 3 mA across the session. This group represents high-frequency stimulation.
  Arms: 100Hz TENS Group
Device: Placebo TENS — Participants use a TENS device identical in appearance to the active treatment units. The power light is on, but no electrical stimulation is delivered due to internal circuit disconnection. Sessions follow the same schedule and duration as the active groups.
  Arms: Placebo TENS Group

SUMMARY:
This study tests whether slow or fast electrical nerve stimulation (TENS) works better to improve arm movement in people recovering from a stroke. Participants will receive TENS on their weak arm three times a week for eight weeks. The results will help find the best TENS setting to support stroke recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 85 years
2. Clinical diagnosis of stroke (ischemic or hemorrhagic) within the past 10 days to 2 months
3. Presence of voluntary movement in the non-paretic arm and at least minimal antigravity movement in the paretic shoulder
4. At least 5 degrees of active wrist extension on the paretic side
5. Able to provide informed consent

Exclusion Criteria:

1. Uncontrolled medical, cardiovascular, or orthopedic conditions
2. Contraindications to TENS (e.g., implanted cardiac pacemaker, skin allergies)
3. Receptive aphasia preventing informed consent or cooperation
4. Significant peripheral neuropathy affecting upper limbs
5. Current participation in another clinical trial or drug study
6. Severe contractures in the shoulder, elbow, wrist, or fingers

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment for Upper Extremity (FMA-UE) | Baseline, Week 4, Week 8, 1-month follow-up, and 3-month follow-up
  Assesses upper limb motor function in stroke patients, including shoulder, elbow, wrist, and hand movements. Scores range from 0 to 66, with higher scores indicating better motor function.

SECONDARY OUTCOMES:
Manual Muscle Testing (MMT) for Wrist Flexion and Extension | Baseline, Week 4, Week 8, 1-month follow-up, 3-month follow-up
  Evaluates muscle strength on a 0-5 scale, where 0 indicates no muscle activity and 5 indicates normal strength.
Modified Ashworth Scale (MAS) for Wrist Flexor Spasticity | Baseline, Week 4, Week 8, 1-month follow-up, 3-month follow-up
  Measures resistance during passive muscle movement on a 0-4 scale to assess spasticity.
Lindmark Motor Score - Grasp Function Subscale | Baseline, Week 4, Week 8, 1-month follow-up, 3-month follow-up
  Assesses hand grasp function on a 0-3 scale based on ability to grip and hold a tennis ball.
Barthel Index | Baseline, Week 4, Week 8, 1-month follow-up, 3-month follow-up
  Evaluates independence in basic activities of daily living. Scores range from 0 to 100, with higher scores indicating greater independence.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuyong People's Hospital, Bao'an District, Shenzhen, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol